CLINICAL TRIAL: NCT00399048
Title: A Randomized, Repeated- Dose, Parallel-Group Comparison of Safety, Efficacy, and Quality of Life Measures With Dilaudid CR (Hydromorphone HCI) or Oxycontin (Oxycodone HCI) in Patients With Chronic Osteoarthritis
Brief Title: An Effectiveness, Safety and Quality of Life Measures With Hydromorphone HCL, Dilaudid CR (Controlled Release)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013270
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Pain; Osteoarthritis; knee Osteoarthritis; hip Osteoarthritis .
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Pain; Osteoarthritis | interventions — Oxycodone

INTERVENTIONS:
Drug: OROS hydromorphone HCL ; OxyContin

SUMMARY:
The purpose of this study was to characterize the effectiveness and safety of OROS hydromorphone HCL and OxyContin in patients with chronic osteoarthritis (OA) of the knee or hip who are receiving chronic nonsteroidal anti-inflammatory drug (NSAID) or other nonsteroidal, non-opioid analgesic (ie, acetaminophen or aspirin) therapy.

DETAILED DESCRIPTION:
This was a multicenter, open-label, randomized (patients are assigned different treatments based on chance), dose-titration, parallel-group study characterizing the effectiveness and safety of OROS hydromorphone HCL and OxyContin in adult patients with osteoarthritis (OA) of the knee or hip who were unable to consistently control or treat their osteoarthritis pain with non opioid medications or with as-needed use of an opioid analgesic. The study consisted of a 14-day period for randomization, dose-titration, and stabilization, followed by a 4-week maintenance phase. Eligible patients were randomized equally to begin therapy with either OROS hydromorphone HCL 8 mg daily or OxyContin 10 mg twice daily. Upward dose titration (doses with increase in titration) from the starting doses was allowed every 2 days, based on pain relief and opioid-related side effects. The dose was to have been titrated to provide the best balance between pain relief and side effects. After 14 days, if therapeutic efficacy with dose stabilization had been documented, the patient was allowed to begin the 4-week maintenance phase. The expected primary efficacy variable endpoints were: The mean pain relief score at endpoint defined as the mean of the last 2 non missing pain relief scores during the Maintenance Phase, and the days from study medication initiation to the third day of moderate to complete pain relief on the patient's final titrated dose (as reported in the patient diary) during the Randomization, Titration and Stabilization Phase. Safety was evaluated by adverse events (AEs), vital signs, and physical examinations. OROS hydromorphone HCL 8mg tablet orally daily or OxyContin 10mg tablet orally daily; Upward dose titration from the starting doses was allowed every 2 days, based on pain relief and opioid-related side effects; After 14 days of efficacy with dose stabilization, patient was allowed to begin the 4 week maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient who met criteria (functional Class I-III in the hip or knee) for osteoarthritis for at least 3 months before enrollment
* Patient who had moderate to severe chronic pain despite regular use and stable doses of an NSAID (nonsteroidal anti-inflammatory drug) or an NSAID with opioid analgesic taken as needed but not on a daily basis for the treatment of osteoarthritis.

Exclusion Criteria:

* Patient intolerant of or hypersensitive to hydromorphone or oxycodone
* Patient of childbearing potential must use medically recognized contraceptive program before and during the study
* Pregnant or breastfeeding
* Patient who had prior joint replacement of the target knee or hip
* Patient with significant respiratory compromise or depressed ventilatory function
* Patient who was known active drug abuser or alcoholics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Two primary efficacy:The mean pain relief score at endpoint during the Maintenance Phase. The day from study medication initiation to the third day of moderate to complete pain relief on the final titrated dose during all three phases.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA